CLINICAL TRIAL: NCT04258462
Title: Hyperpolarized 13C Pyruvate Metabolic MRI to Predict Renal Tumor Aggressiveness
Brief Title: Hyperpolarized 13C Pyruvate MRI Scan in Predicting Tumor Aggressiveness in Patients With Renal Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhen Wang, MD (Other)
Collaborators: American Cancer Society, Inc. (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Zhen Wang, MD, Professor of Radiology, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18525; NCI-2018-03692 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R01CA249909 (NIH)
Record Dates: First submitted 2019-09-02; First posted 2020-02-06 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Benign Kidney Neoplasm; Kidney Neoplasm; Renal Cell Cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diagnostic (HP 13C pyruvate with MRI) (Experimental): Participants receive HP 13C pyruvate IV and then undergo 13C MRI scan 1-2 minutes post HP 13C pyruvate injection. Participants may receive an optional second HP 13C pyruvate injection and undergo 13C pyruvate MRI scan 15 to 30 minutes following completion of the first scan or at a return visit 1-2 weeks from the first HP C13 MRI
  Interventions: Drug: Hyperpolarized Carbon C 13 Pyruvate; Procedure: Magnetic Resonance Imaging
- Diagnostic (Combined (co-polarized) HP 13C pyruvate and 13C, 15N2 Urea with MRI) (Experimental): Participants receive HP 13C pyruvate and 13C 15N2 urea IV and then undergo an MRI scan 1-2 minutes post injection. Participants may receive an optional second HP 13C pyruvate with 13C 15N2 urea injection and undergo a second MRI scan 15 to 30 minutes following completion of the first scan or at a return visit 1-2 weeks from the first HP C13 MRI
  Interventions: Drug: Hyperpolarized Carbon C 13 Pyruvate; Procedure: Magnetic Resonance Imaging; Drug: Hyperpolarized 13C,15N2-urea

INTERVENTIONS:
Drug: Hyperpolarized Carbon C 13 Pyruvate — Given IV
  Other Names: Hyperpolarized 13C-Pyruvate; Hyperpolarized Pyruvate (13C)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MRI; MRI Scan; Nuclear Magnetic Resonance Imaging
Drug: Hyperpolarized 13C,15N2-urea — Given IV
  Other Names: HP 13C, 15N2
  Arms: Diagnostic (Combined (co-polarized) HP 13C pyruvate and 13C, 15N2 Urea with MRI)

SUMMARY:
This feasibility study will evaluate how well hyperpolarized 13C pyruvate magnetic resonance imaging (MRI) scan works in predicting tumor aggressiveness in participants with renal tumors. Hyperpolarized 13C pyruvate is a non-radioactive substance with potential usage in the diagnostic imaging of tumors. Hyperpolarized 13C pyruvate MRI may help doctors determine non-invasively whether a kidney tumor is a benign tumor or cancer, and if cancer, how aggressive it is. This may help doctors and participants with renal tumors in the future to make better treatment decisions.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

1. To investigate the association between HP 13C pyruvate-to-lactate conversion (peak lactate/pyruvate ratio, lactate /pyruvate AUC (area under the curve), the apparent rate constant (kPL) and renal tumor histology (benign renal tumors versus RCCs) and grade (low vs high grade in cases of RCCs).

SECONDARY OBJECTIVES:

1. To determine the reproducibility of HP 13C pyruvate MRI in participants who undergo an optional second HP 13C pyruvate MRI.
2. To investigate the association between HP 13 C pyruvate-to-lactate conversion and tumor growth rate in participants who are deemed clinically appropriate for active surveillance for their renal tumors.
3. To determine the safety of HP 13C pyruvate in renal tumor participants.

EXPLORATORY OBJECTIVES:

1. To investigate the association between HP markers (peak lactate/pyruvate, lactate /pyruvate AUC, kPL) and tissue-based markers including Lactate Dehydrogenase A (LDHA) expression and lactate dehydrogenase (LDH) activity, and Monocarboxylate transporter 4 (MCT4) expression on tumor tissues from surgical specimen or from biopsy.
2. To explore the correlation between HP 13C pyruvate-to-lactate conversion (peak lactate/pyruvate ratio, lactate/pyruvate AUC (area under the curve), the apparent rate constant kPL) and 13C urea tissue perfusion in the kidneys and renal tumors.

OUTLINE:

Participants receive HP 13C pyruvate intravenously (IV) or a combination of co-polarized 13C pyruvate and 13C, 15N2 Labeled urea (15N2) and then undergo MRI scan 1-2 minutes post injection

Participants may receive an optional second HP 13C pyruvate intravenously (IV) or a combination of hyperpolarized 13C pyruvate and 13C, 15N2 urea injection and undergo 13C pyruvate MRI scan 15 to 30 minutes following completion of the first scan during the same imaging session, or the participant can return for a separate visit within 1-2 weeks from the first MRI to receive the optional second scan.

After completion of study treatment, participants are followed up 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Renal tumor measuring 1 cm and greater in diameter. To minimize any potential partial volume effects in this pilot study, the investigators have limited the lower size range of the tumor to 1 cm. The investigators will include all renal tumor measuring 1 cm and greater in diameter in this first study to facilitate obtaining tumors of a range of histology and grade.
2. The participant is being considered by the treating physician to have any of the following management options: partial or radical nephrectomy, ablation, or active surveillance for his/her renal tumor.
3. The participant is able and willing to comply with study procedures and provide signed and dated informed consent.
4. The participant is willing to undergo standard of care abdominal MRI in connection with the study exam.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Exclusion Criteria:

1. Participants who because of age, general medical or psychiatric condition, or physiologic status cannot give valid informed consent.
2. Participants unwilling or unable to undergo magnetic resonance (MR) imaging, including patients with contra-indications to MR imaging, such as cardiac pacemakers or non-compatible intracranial vascular clips.
3. Any metallic implant or device that distorts local magnetic field and compromises the quality of MR imaging of the abdomen.
4. Prior focal therapy (i.e. ablation) for the renal tumor.
5. Poorly controlled hypertension, with blood pressure at study entry >160/100. The addition of anti-hypertensives to control blood pressure is allowed for eligibility determination.
6. Congestive heart failure or New York Heart Association (NYHA) status >= 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison between HP 13C pyruvate-to-lactate conversion, as measured by peak lactate/pyruvate ratio with tumor histology and grade. | Up to 12 months
  Descriptive statistics (mean, median, standard deviation, distribution, etc) of the metabolism measures will be calculated. The investigators will use a tree-based cross-validated Classification & Regression Trees (CART) model for predicting benign renal tumors vs. low grade renal cell carcinoma (RCC) vs. high grade RCCs based on the HP 13C pyruvate metabolic data
Comparison between HP 13C pyruvate-to-lactate conversion, as measured by the lactate /pyruvate area under curve (AUC) with tumor histology and grade. | Up to 12 months
  Descriptive statistics (mean, median, standard deviation, distribution, etc) of the metabolism measures will be calculated. We will use a tree-based cross-validated Classification & Regression Trees (CART) model for predicting benign renal tumors vs. low grade RCCs vs. high grade RCCs based on the HP 13C pyruvate metabolic data;
Comparison between HP 13C pyruvate-to-lactate conversion, as measured by the apparent rate of constant metabolic flux of HP 13C-pyruvate to lactate (kPL), with tumor histology and grade. | Up to 12 months
  Descriptive statistics (mean, median, standard deviation, distribution, etc) of the metabolism measures will be calculated. The investigators will use a tree-based cross-validated Classification & Regression Trees (CART) model for predicting benign renal tumors vs. low grade RCCs vs. high grade RCCs based on the HP 13C pyruvate metabolic data;

SECONDARY OUTCOMES:
Estimate of intra-subject agreement for those with optional second scan | Up to 12 months
  For participants who obtained an optional second HP 13 C pyruvate magnetic resonance imaging (MRI), intraclass correlation coefficient (ICC) will be used to estimate the intra-subject agreement. ICCs will be obtained from a one-way analysis of variance model based on 2 serial measurements per subject. The ICC ranges from 0 to 1. An ICC close to 1 indicates high similarity between values from the same group. An ICC close to zero means that values from the same group are not similar. The results will be presented with a 95% confidence interval.
Comparison of the HP 13C metabolism measures to change in tumor size | Up to 12 months
  For participants who are in active surveillance for their renal tumors, MRI findings will be compared to tumor growth rate while on active surveillance. Correlations of HP 13C metabolism measures to change in tumor size on subsequent surveillance imaging studies will be performed using Pearson or rank correlation.
Incidence of treatment-related adverse events | 1 day, 30 minutes following hyperpolarized 13C pyruvate injection
  Assessment of the occurrence of clinically significant changes in safety variables from baseline. Safety endpoints include monitoring for the occurrence of treatment-emergent AEs. Toxicities will be graded using the National Cancer Institute (NCI) Common Terminology (Toxicity) Criteria for Adverse Events (CTCAE) version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Jane Wang, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-06-13): https://cdn.clinicaltrials.gov/large-docs/62/NCT04258462/ICF_000.pdf